CLINICAL TRIAL: NCT04487548
Title: Perioperative Smoking Cessation BUndle in a Tertiary Care Hospital - Can Turning Virtual Improve Outcomes? A Pilot Randomized Controlled Trial.
Brief Title: Perioperative Smoking Cessation BUndle in a Tertiary Care Hospital - Can Turning Virtual Improve Outcomes?
Acronym: BuTT-Out
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: Royal Columbian Hospital Foundation (Other)
Responsible Party: Principal Investigator, Susan Lee, Physician, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FHREB 2017-099
Record Dates: First submitted 2018-03-16; First posted 2020-07-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-09

CONDITIONS: Smoking Cessation; Surgical Complications
Keywords: Smoking; Surgery; Anesthesia; Complications
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Intervention Model Description: Study Design This pilot randomized controlled trial with two parallel arms will be undertaken with current smokers who are scheduled for elective surgery at RCH. Participants will be randomized to a smoking cessation bundle (video, electronic or mailed brochure, referral to QuitNow.ca Smokers' Helpline and pharmacological smoking cessation therapy) or standard care (advice to quit and inconsistent recommendation of resources).
  All current adult smokers being scheduled for elective surgery at RCH will be invited to participate. The investigators plan on recruiting 30 participants with 15 participants per group. Every eligible patient will be invited to participate.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Blinding of study participants is not possible. Blinding of staff may not always be possible, although staff will not be informed which group the participant has been randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The control group will have their preadmission clinic telephone call as normal and may be given advice to quit smoking and information about available smoking cessation resources over the phone.
- Intervention group (Experimental): The intervention group will be emailed (or postal mailed) the smoking cessation bundle with educational video, brochure, referral to the Smokers' Helpline and direct referral to an online pharmacy for nicotine replacement.
  Interventions: Other: Remote smoking cessation bundle

INTERVENTIONS:
Other: Remote smoking cessation bundle — The bundle is a remote version of what has previously been described in prior literature, which includes:
  1. A brief (<5 minutes) advice
  2. Preoperative smoking cessation video prepared by QuitNow
  3. Patients will be provided brochures on smoking cessation
  4. A referral will be faxed (or internet-registered) to the Quitnow.ca Smokers' Helpline
  5. All patients will be requested to participate in the provincial Smoking Cessation program that provides a free 12-week supply of NRT once per year.
  Arms: Intervention group

SUMMARY:
Smoking continues to be a burden to the healthcare system in Canada. It is well-known that smokers suffer more complications and higher risk of mortality after surgery than non-smokers. A quality improvement project at Royal Columbian Hospital recently showed that it is possible to implement a smoking cessation bundle for all current smokers during their preadmission clinic visit. However, due to the COVID-19 pandemic, much of the bundle was abandoned as it relied heavily on in-person interactions. The investigators wish to study the effect of a structured smoking cessation bundle, delivered remotely, on smoking cessation and postoperative complications. The aim is to determine the feasibility of giving the remotely delivered bundle to elective surgical patients before or around the time of a preadmission clinic visit, and whether it can reduce smoking rates and postoperative complications versus the standard uncoordinated advice.

DETAILED DESCRIPTION:
Introduction and Background Smoking continues to be a burden to the healthcare system in Canada. As of 2019, 3.7 million Canadians (12% of the population over age 15) reported being a current smoker. British Columbia's smoking rate is lower, but 10.2% of adults still regularly smoke cigarettes1. It is well-known that smokers suffer more complications and higher risk of mortality after surgery than non-smokers. Pulmonary complications, cardiovascular complications, and surgical site infections are mediators of smoking-associated mortality at 6-months and 1-year after elective surgery.

Although there have been a handful of studies that have demonstrated dramatic reductions in postoperative complications with well-timed smoking cessation interventions in the preoperative period, these results have not translated into widespread clinical practice in delaying surgery for the purpose of achieving smoking cessation. In addition, most of these studies took place in Europe, where smokers may behave differently than in the Canadian setting.

A systematic review recommended at least 4 weeks of smoking cessation in order to reduce postoperative complications6. Several European studies have shown dramatic reductions in complications (up to 30% absolute risk reductions) when smoking cessation interventions have been implemented 4-8 weeks preoperatively. One Canadian editorial even suggested new policies be put into place to delay elective surgeries in smokers until a trial of cessation for 6 weeks had taken place.

Implementation of smoking cessation programs preoperatively have the potential to reduce morbidity and mortality. A Cochrane systematic review has shown that preoperative smoking cessation therapy improves both short and long-term smoking cessation. In fact, a surgical encounter with the healthcare system has been described as a "teachable moment" that provides motivation for patients to permanently stop smoking. Despite this information, most anesthesiologists do not routinely offer smoking cessation advice to their patients and advice, counselling, and pharmacotherapy for smoking cessation is not routine in pre-admission clinics across Canada and the United States.

Several small trials have shown that smoking cessation interventions can increase smoking cessation and reduce postoperative complications, particularly wound-healing complications, which can have an absolute risk reduction of up to 25%. Prior work by one of the co-investigators showed that a simple intervention in the pre-admission clinic was able to increase the abstinence rate from 3.6% to 14.3% on the day of surgery. Smoking cessation initiated in the perioperative period can also promote long-term smoking cessation.

Despite these successes, since the COVID-19 pandemic, standard care at Royal Columbian Hospital (RCH) has not routinely included specific preoperative smoking cessation pharmacotherapy or counselling. However, hospital leaders and the RCH Department of Anesthesia have identified preoperative preparation, including smoking cessation, as a key area of interest for development. Therefore, this is the ideal time to study the feasibility of the perioperative smoking cessation bundle given to patients without the requirement for an in-person visit. Advantages of this remote model are expected to continue after the pandemic restrictions end, since smoking cessation bundles will be able to be started earlier (and thus have more potential to prevent surgical complications), compared to waiting for a preadmission clinic visit, which can often occur only a few days preoperatively. The perioperative smoking cessation bundle will include: an emailed link to a quitnow.ca preoperative smoking cessation video and referral to quit coach, free nicotine replacement therapy (NRT) delivered by an online pharmacy, an emailed or post-mailed RCH smoking cessation brochure, and brief telephone advice. This bundle will be offered to those regular smokers of cigarettes randomized to the intervention group following their surgical consultation, at the time of preadmission clinic appointment booking, or following their preadmission telephone consultation. The control group will receive the standard of care which sometimes includes brief advice and informing patients about availability of further aids.

Once the simple smoking cessation intervention has been implemented for the intervention group, the investigators wish to compare rates of resource access, smoking cessation, and postoperative complications between the group receiving the smoking cessation bundle and those receiving standard care. Due to the COVID-19 pandemic, in-person preadmission clinic visits are no longer scheduled. Instead, high-risk surgical patients are phoned prior to surgery to mitigate surgical risk factors and better prepare them for surgery. Self-identification as a regular smoker is one risk factor that would warrant recruitment into the study.

The investigators estimated that a definitive randomized controlled trial would require a sample size of 214 participants. However, relatively low rates of smoking in British Columbia and the cancellation of in-person preadmission clinic visits present a unique challenge to patient recruitment. It is therefore imperative to establish the recruitment rate for progression to a full randomized controlled trial.

Additionally, a preliminary analysis of rates of smoking and reduction of postoperative complications in elective surgical patients when the smoking cessation bundle is given to patients immediately following their preadmission clinic telephone consultation will be conducted. The investigators plan to carry out a pilot randomized controlled trial where patients who identify as smokers will be randomized to receive the remotely delivered smoking cessation bundle versus standard care.

Purpose and Justification Most randomized studies showing improved smoking cessation rates after preoperative interventions have strict inclusion and exclusion criteria, and required ongoing consent for research experimentation, which limits their external generalizability. The BuTT Out Pilot Study is of utmost importance since it has the potential to demonstrate reductions in surgical site infections and lengths-of-stay using a low-cost intervention (a bundle of emailed video, brochure, helpline referral and government funded smoking-cessation therapy). A 2020 survey of the BC Smoking Cessation Program reported that 66% of respondents found the program helpful, with a quit rate of 37%. Providing the program as a part of a structured bundle will improve the accessibility of smoking cessation aids. If this hypothesis is confirmed as suspected since it is based on prior research in other countries, widespread implementation could translate into tremendous advantages for the patient, in terms of reduced complications, and providers, in terms of cost savings. Conducting a pilot study will help mitigate the challenge of recruiting an adequate sample size by establishing a recruitment rate and consequently improve the feasibility of a definitive randomized controlled trial. Since this study will examine remotely-delivered interventions, its potential for widespread use will be much greater than other previously studied in-person study designs.

Research Question For patients who smoke undergoing elective surgery, what is the effect of an evidence-based remotely-delivered smoking cessation bundle administered preoperatively on patients' outcomes (smoking rates, complication rates and hospital length of stay) compared with standard practice which sometimes includes brief advice and informing patients about availability of further aids?

Research Objectives To establish the recruitment rate, optimal recruitment pathway, and rate of accessing of available resources as criteria for progression to a definitive randomized controlled trial.

To determine whether smoking rates, surgical complications, and postoperative complications can be documented in elective surgical patients when the remotely-delivered smoking cessation bundle is administered preoperatively vs. standard care.

Research Hypothesis The hypothesis for this pilot RCT is that at least 8 patients will be screened per week, at least 25% will give informed consent, and >80% will adhere to the study protocol.

The overarching research hypothesis is that in patients who smoke, receiving the remotely-delivered perioperative smoking cessation bundle prior to elective surgery for the purpose of quitting smoking will result in reduced smoking rates on the day of surgery, lower 30-day complications, and shorter lengths of stay. Definitive estimation of effect size is not expected from this pilot study, but confidence intervals will give rise to sample size estimation for a future full-size trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and over.
2. Current smoker (self-identified from pre-surgical package).
3. Surgery date over 1 week away or not yet booked.

Exclusion criteria

1. Emergency surgery.
2. Smokers who only consume non-cigarette forms of tobacco (pipe, smokeless tobacco).
3. Smokers who only consume marijuana or vaping.
4. Patients who are pregnant or breastfeeding.
5. Inability to provide informed consent.
6. Currently enrolled in any other research study involving smoking cessation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Uptake of smoking cessation resources | Day of surgery
  The primary outcome is the participant's self-reported rate of uptake of smoking cessation information and accessing available resources. Uptake will be assessed by a brief questionnaire given at each of the follow-up time points asking which resources were accessed and if NRT was used.
Uptake of smoking cessation resources | 30 days postoperatively
  The primary outcome is the participant's self-reported rate of uptake of smoking cessation information and accessing available resources. Uptake will be assessed by a brief questionnaire given at each of the follow-up time points asking which resources were accessed and if NRT was used.
Uptake of smoking cessation resources | 8 weeks post-randomization
  The primary outcome is the participant's self-reported rate of uptake of smoking cessation information and accessing available resources. Uptake will be assessed by a brief questionnaire given at each of the follow-up time points asking which resources were accessed and if NRT was used.
Uptake of smoking cessation resources | 6 months postoperatively
  The primary outcome is the participant's self-reported rate of uptake of smoking cessation information and accessing available resources. Uptake will be assessed by a brief questionnaire given at each of the follow-up time points asking which resources were accessed and if NRT was used.

SECONDARY OUTCOMES:
Recruitment rate | Enrollment
  Number of eligible patients consented out of all eligible patients
Recruitment timing | Enrollment
  Duration between enrollment and day of surgery
Participant satisfaction with smoking cessation bundle assessed by study questionnaire | 8 weeks post-randomization
  Open-ended questions asking how satisfied participants were with the smoking cessation bundle, which parts of the bundle were most and least helpful
Change in smoking status from baseline | Day of surgery, 30 days postoperatively, 8 weeks post-randomization and 6 months postoperatively
  Self-report of smoking status at each time point compared to baseline (defined as number of cigarettes smoked in the last 24 hours)
Hospital Length of Stay | First 30 days
  Length of time the participant is admitted to the hospital for their surgical procedure.
Postop complications (day 3 POMS) | Postop Day 3
  Day 3 Postoperative Morbidity Survey (POMS).
Cost of nicotine replacement therapy | 6 months
  Total cost of NRT prescriptions supplied
Number of nicotine replacement therapy refills | 6 months
  For those using NRT, how many times did they refill their NRT prescription
Number of nicotine replacement therapy pharmacy deliveries | 6 months
  For those using NRT, how many pharmacy deliveries of NRT did they get

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Lee, MD, FRCPC, Principal Investigator — Fraser Health Authority; Michelle Mozel, MSc, Study Chair — Fraser Health Authority
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pillar M, Sara R, Burditt D, Rai RK, Monteiro L, Lertnamvongwan R, Mozel M, Merchant R, Lee SM. A pilot randomized trial of a virtual perioperative smoking cessation bundle in a tertiary care hospital. Can J Surg. 2025 Nov 13;68(6):E460-E468. doi: 10.1503/cjs.016224. Print 2025 Nov-Dec. PMID 41233153